CLINICAL TRIAL: NCT06445777
Title: Impact of Preventive Mental Health Programme on Social/Emotional Functioning and Resilience in Children in South Africa
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Little Lions Child Coaching (Other)
Collaborators: University of Cape Town (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: LLRCT
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Psychological Well-Being
Keywords: Emotional Resilience; Mental Health Prevention; South Africa; Universal Mental Health Promotion
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Children will be randomly assigned to either the control or intervention group after the baseline assessment. Participants in the control group will receive the intervention at a later stage.
Who Masked: Investigator
Masking Description: The researchers involved in data collection after the intervention will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Behavioural/ psychosocial intervention (i.e., mental health prevention and promotion programme) to boost emotional awareness, confidence, coping skills, and resilience.
  Interventions: Behavioral: Mental Health Prevention and Promotion
- Control Group (No Intervention): Participants in the control group will receive the intervention at a later stage.

INTERVENTIONS:
Behavioral: Mental Health Prevention and Promotion — The Inner Lion Programme is made up of 12 interactive workshops which are based on four key pillars: building confidence by identifying strengths and personal qualities; improving emotional intelligence and self-awareness; establishing adaptive coping strategies and channels of support; and boosting resilience. Professionally created by Child Psychologist Stijn de Leeuw together with an advisory team of psychologists from the Netherlands and South Africa, the programme follows a carefully structured and curated prevention and promotion mental health curriculum with games, crafting activities, psycho-educational stories, dance, movement, and breathing exercises. Workshops are led by local role models (a male-female duo) with lived experience trained to be mental health coaches.
  Other Names: Inner Lion Programme
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to test the effectiveness of a mental health prevention and promotion programme delivered to children (ages 8 to 13) living in under-resourced communities in South Africa.

The main question it aims to answer is:

Does the programme increase resilience and improve psychological well-being?

Participants will be asked to attend the programme twice a week after school for a period of six weeks and complete a series of questionnaires.

Researchers will compare children who attended the programme to those who did not to see if the programme resulted in better social/emotional functioning and resilience.

DETAILED DESCRIPTION:
Although the well-being of vulnerable South African children is a significant public health concern, few studies have evaluated the effectiveness of mental health prevention and promotion interventions in low- and middle- income countries. Little Lions Child Coaching is a South African youth-led, community-based non-governmental organisation (NGO) that aims to normalise mental health conversations and empower the next generation to tap into their emotional resilience by providing accessible mental health support to children in under-resourced communities surrounding Cape Town.

The aim of this effectiveness study is to measure how a mental health prevention and promotion programme, designed and implemented by Little Lions Child Coaching, impacts the resilience and social/emotional functioning of children (ages 8 to 13) living in townships surrounding Cape Town.

Participants in the intervention condition will receive the programme twice a week after school for a period of six weeks to boost their emotional awareness, confidence, coping skills and resilience. Resilience scores will be compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Between 8 and 13 years old
* Fluent in Xhosa and/or English
* Lives in one of the following communities in Cape Town, South Africa: Khayelitsha, Langa, or Mfuleni

Exclusion Criteria:

* Younger than 8 years old or older than 13 years old
* Do not have a strong understanding of the language of instruction (i.e., Xhosa/English)
* Lives in an area outside of Khayelitsha, Langa, or Mfuleni

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in resilience scores using the Child and Youth Resilience Measure | At baseline and in 6 weeks
  Higher scores on the Child and Youth Resilience Measure indicate greater resilience. The minimum score is 17 and the maximum score is 51. A t-test will be used to determine whether the control versus intervention group had significantly different mean scores on the Child and Youth Resilience measure after the intervention relative to the baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Malcolm-Smith, Principal Investigator — University of Cape Town
Locations (1):
- Neighbourgood, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with an academic interest in the effectiveness of universal mental health interventions for children and adolescents. To protect personal information, all data shared will be coded.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact caitlin@littlelionschildcoaching.com